CLINICAL TRIAL: NCT02858336
Title: CaREFREE Study (Calorie Restriction, Environment and Fitness: Reproductive Effects Evaluation Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 160157; 16-E-0157
Record Dates: First submitted 2016-08-05; First posted 2016-08-08 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-06-09

CONDITIONS: Hormones
Keywords: Luteinizing Hormone (LH); Weight Loss; Functional Hypothalamic Amenorrhea (HA); Gonadotropin-Releasing Hormone (GnRH); Energy Deficiency
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): All participants will receive the NEA availability to act as their own control to the experimental DEA intervention.
  Interventions: Behavioral: NEA
- Experimental (Experimental): All participants will be in the experimental arm and receive the DEA intervention.
  Interventions: Behavioral: DEA

INTERVENTIONS:
Behavioral: NEA — Neutral Energy Availability: 5-day outpatient intervention of prescribed diet and exercise to elicit an energy availability of 45 kcal/kg LBM day.
  Arms: Control
Behavioral: DEA — Deficient Energy Availability: 5-day outpatient intervention of prescribed diet and exercise to elicit an energy availability of 20 kcal/kg LBM day.
  Arms: Experimental

SUMMARY:
Background:

Functional hypothalamic amenorrhea (functional HA) is a condition where a woman s period stops for a temporary time. This is due to improper function of the hypothalamus. This is the part of the brain that directs the whole reproductive system. Researchers want to learn more about functional HA. They also want to learn how diet, exercise, and other factors may change women s menstrual cycles.

Objective:

To better understand functional HA.

Eligibility:

Healthy women ages 18-28 years old who:

* Have regular periods
* Exercise no more than 4 hours a week
* Had their first period at age 11-14

Design:

Participants will be prescreened over the phone.

Participants will be screened with:

* Blood and urine tests
* Medical history
* Physical exam.

Participants will have 9 or 10 visits over about 3 menstrual cycles. These include:

* Repeat of screening tests
* Questionnaires
* Exercise test
* Resting energy expenditure test: Participants fast overnight before the test. They lie on their back under a canopy for a half hour.
* Body composition test: This is done with a dual energy x-ray absorptiometry (DXA) scan.
* Pelvic ultrasound
* For two full-day visits, an IV is inserted into an arm vein. The IV takes a blood sample every 10 minutes for 8 hours.

Participants will keep logs:

* Menstrual cycle log
* Diet log for three 4-day cycles

Participants will receive test kits to complete at home:

* Daily blood and urine sample
* Ovulation

Participants will take a daily iron supplement. They will wear a wristband that monitors activity 24 hours a day.

Participants will stick to a special diet for two 5-day periods of time. They will complete two 4-day exercise programs.

DETAILED DESCRIPTION:
Functional hypothalamic amenorrhea (HA) is a reversible form of hypogonadotropic hypogonadism (HH) that can be triggered by stressors such as exercise, nutritional deficits, and psychological stress. Dysfunction of the hypothalamic component of the reproductive axis plays a key role in functional HA and is manifest by an altered pattern of luteinizing hormone (LH) pulses detectable in peripheral blood. There is ample evidence supporting the use of LH as a surrogate marker of hypothalamic gonadotropin-releasing hormone (GnRH) secretion from the hypothalamus. There is also significant evidence that women vary in their susceptibility to such stress-induced amenorrhea, pointing to a role for both environmental and genetic factors in the etiology of functional HA. However, the variation in changes in GnRH pulse frequency in response to stressors in healthy women has not been defined. Data from previous work in our lab has suggested that rare variants in genes associated with other forms of HH may also contribute to the variability seen in susceptibility to functional HA. The long-term goal of our research is to examine the interaction of environment and genes in HA. In this pilot study we propose to examine the inter-individual variability in pulsatile LH secretion in response to standardized neutral and deficient energy availability (NEA and DEA, respectively) in normal women. We will then relate this primary end-point to proposed predictive factors including past reproductive and family history and markers of current metabolic status and their response to energy availability. Our initial analyses will help to determine simplified biomarkers that can be translated to larger studies examining the potential combined effect of energy availability and genotype.

The proposed pilot study is a single-site, 2-period study in healthy female volunteers. The study will enroll approximately 300 participants with a target for study completion of 36 subjects. Eligible participants will be females >= 18 years of age. Eligible participants will have had menarche at or before 14 years of age and no earlier than age 11. Eligible participants will have a gynecological age (years after menarche) of 14 years or less. The upper age limit will vary based on each subject s age of menarche and fall between 25 and 28 among participants. Eligible participants will confirm at the pre-screening call having normal menstrual cycles (self-reported) for at least the previous 2 months and ovulation will be confirmed during the menstrual cycle before the start of intervention.

The primary outcome will be changes in daytime LH pulse frequency, when comparing NEA vs DEA. Secondary measures will evaluate past reproductive history, family history, and current metabolic status using medical history interviews, lifestyle questionnaires and maximum oxygen uptake (as a measure of fitness). Resting energy expenditure, body composition as well as metabolic and stress hormones will be measured at baseline and in association with the interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be enrolled with distribution across race. Each potential participant must meet all of the following inclusion criteria in order to be eligible to enroll in the study:

1. Female
2. Between 18 and 28 years of age (inclusive)
3. Reported menarche between the ages of 11 and 14 years
4. Gynecological age of <= 14 years
5. A history of self-reported regular menstrual cycles when not on contraceptive medication of between 25 and 35 days (inclusive) at prescreen and knowledge of date of onset of menses before the screening visit
6. A BMI of 18.5 to 27 kg x m^2 and a weight >= 93 lbs.
7. Agrees to use barrier contraception method for the duration of the study and the follow up period
8. Agrees to abstain from alcohol consumption during both 5-day diet/exercise study interventions
9. Agrees to abstain from donating blood during the study and within 30 days of completing the study
10. Agrees to abstain from biotin supplements for the duration of the study
11. Is willing and able to fulfill the requirements of the protocol and to provide informed consent
12. Able to speak and read English
13. Lives within 50 miles of the Clinical Research Unit

EXCLUSION CRITERIA:

A potential participant meeting any of the following exclusion criteria is not eligible to enroll in the study:

1. Currently lactating or pregnant or planning on becoming pregnant for the duration of the study
2. Has ever given birth
3. History in the past 3 months of dieting or weight loss amounting to greater than 2 kg
4. > 4 hours per week of aerobic exercise for the past 3 months
5. Has initiated training for an athletic sport or event in the past 3 months that, in the opinion of the investigator, may interfere with the results of the study
6. Currently using hormone-based contraception, including those administered orally, vaginally, via injection, sub-dermally, or transdermally
7. Current use of medications or supplements that may interfere with the results of the study, including:

   i.Steroids

   ii.Hormone-based contraception

   iii.Sleeping pills

   iv.Homeopathic substances (e.g. Chinese herbs, protein or other powders, and other-the-counter extracts)

   v.Stimulants (e.g. Ritalin)

   vi.Antidepressants or anti-epileptic medications or centrally acting anti-hypertensive medications
8. Current use of recreational drugs (alcohol intake will be monitored and excluded during the two intervention periods)
9. Unable to consume food containing dairy or nuts
10. Has regular overnight awake periods, for example overnight or rotating shift work, that will continue during the study, at the discretion of the investigator
11. Has currently or has a history of any of the following: autoimmune, heart, liver, renal disease, diabetes, or another health condition deemed by the PI to be a contraindication to study participation.

Additional Eligibility Criteria to be Met Prior to Start of Intervention(s):

Criteria 1 Habitual energy intake between 35-55 kcal/kg LBM*day

Criteria 2 VO2max <= 40 ml/kg/min with the option to increase this at the discretion of the PI, depending on the current and past exercise level of the participant.

Criteria 3 Hemoglobin, prolactin and TSH within normal female range for testing laboratory.

Criteria 4 Ovulation confirmed in the cycle before each study intervention by self-reported positive urine test, ultrasound and/or progesterone blood-levels

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be change in daytime LH pulse frequency following 5 days of neutral energy availability as compared to LH pulse frequency following 5 days deficient energy availability. LH pulse frequency. | NEA Intervention Day 5 and DEA Intervention Day 5
  Change in LH pulse frequency collected by sampling every 10 minutes over 8 hours during a study visit.

SECONDARY OUTCOMES:
Change in hormone measures (LH, FSH, estradiol, and progesterone) from daily urine samples and blood spots, total cycle, follicular and luteal phase length during the cycle following NEA or DEA | Menstrual cycle of the NEA Intervention and menstrual cycle of DEA Intervention
  Change in Laboratory Values during each menstrual cycle.
Change in leptin, ghrelin, adiponectin, insulin, and glucose in response to standardized breakfast, lunch, and snack | NEA Intervention Day 5 and DEA Intervention Day 5
  Change in Laboratory Values collected by sampling after standardized breakfast, lunch, and snack over 8 hours during a study visit.
Change in cortisol, TSH, TT3, and fT4 | NEA Intervention Day 5 and DEA Intervention Day 5
  Change in Laboratory Values collected by sampling over 8 hours during a study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie D Shaw, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We intend to make individual participant data available through collaboration or upon reasonable request.

REFERENCES:
- [Background] Loucks AB. The response of luteinizing hormone pulsatility to 5 days of low energy availability disappears by 14 years of gynecological age. J Clin Endocrinol Metab. 2006 Aug;91(8):3158-64. doi: 10.1210/jc.2006-0570. Epub 2006 May 23. PMID 16720651
- [Background] Loucks AB, Thuma JR. Luteinizing hormone pulsatility is disrupted at a threshold of energy availability in regularly menstruating women. J Clin Endocrinol Metab. 2003 Jan;88(1):297-311. doi: 10.1210/jc.2002-020369. PMID 12519869
- [Background] Williams NI, Young JC, McArthur JW, Bullen B, Skrinar GS, Turnbull B. Strenuous exercise with caloric restriction: effect on luteinizing hormone secretion. Med Sci Sports Exerc. 1995 Oct;27(10):1390-8. PMID 8531610
- [Derived] Shekhar S, Tessa Tonleu J, Okigbo CC, Leka H, Kim AE, Purse BP, Hirsch KR, Stolze BR, McGrath JA, Smith-Ryan AE, Soldin SJ, Hall JE. Thyroid axis adaptations to moderate short-term energy restriction in healthy, young women. Eur J Endocrinol. 2025 Apr 30;192(5):568-576. doi: 10.1093/ejendo/lvaf083. PMID 40265345
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-E-0157.html